CLINICAL TRIAL: NCT04590365
Title: Efficacy of Carrageenan Nasal and Throat Spray for COVID-19 Prophylaxis - A Double Blind Randomised Placebo-controlled Trial
Brief Title: Carrageenan Nasal Spray for COVID-19 Prophylaxis
Acronym: ICE-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Cardiff University (Other); Marinomed Biotech AG (Industry); Walgreens Boots Alliance (Other); Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 283187
Record Dates: First submitted 2020-05-28; First posted 2020-10-19 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: Carrageenan; Nasal spray; Anti-viral; Prevention; Carragelose
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study design consists of a double blind, randomised placebo-controlled trial. Of the 480 participants recruited, 240 participants will be randomly allocated to each of either the treatment arm (verum Coldamaris plus i.e. Iota-Carrageenan 0.12% plus 0.04% Kappa-Carrageenan in 0.5% saline) or placebo (Coldamaris sine i.e. 0.5% saline) arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation to each group, treatment or placebo administration and data analysis will be blinded to both participant and investigator. The sprays will be blinded at the site of manufacture. Trial sealed envelopes will be available in case of any adverse reactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coldamaris plus (Experimental): verum Coldamaris plus i.e. 0.12% Iota-Carrageenan plus 0.04% Kappa-Carrageenan in 0.5% saline
  Interventions: Device: Carrageenan nasal and throat spray
- Coldamaris sine (Placebo Comparator): Coldamaris sine i.e. 0.5% saline
  Interventions: Device: Saline nasal and throat spray

INTERVENTIONS:
Device: Carrageenan nasal and throat spray — Iota-carrageenan nasal and throat spray (verum Coldamaris plus i.e. Iota-Carrageenan 0.12% plus 0.04% Kappa-Carrageenan in 0.5% saline)
  Arms: Coldamaris plus
Device: Saline nasal and throat spray — Saline nasal and throat spray (placebo Coldamaris sine i.e. 0.5% saline)
  Arms: Coldamaris sine

SUMMARY:
The current COVID-19 pandemic is the biggest global healthcare challenge in the last century, and the number of cases in the next 12 months is likely to increase. There is currently no proven treatment, chemoprophylaxis or vaccine against COVID-19, which exhibits a wide clinical spectrum from asymptomatic carriage to mild upper respiratory tract infection, severe viral pneumonia to acute respiratory distress syndrome and death. Key workers are at high risk of exposure highlighting the need for effective preventative strategies.

SARS-CoV-2 is a positive-sense single-stranded enveloped RNA virus which transmits via droplets, aerosols and direct contact, to reach their target naso- and oropharyngeal epithelial cells through initial electrostatic interactions to cell surface heparan sulphate (HS) proteoglycans. Carrageenan mimics cell surface HS, thereby trapping the virus to allow mucociliary clearance and has demonstrated anti-viral activity in-vitro and in a number of common cold clinical trials when administered as a nasal spray.

ICE-COVID a randomised, double blind, placebo-controlled phase III trial of the prophylactic efficacy of iota-carrageenan nasal and throat spray in preventing COVID-19 illness in at risk healthcare professionals. Participants (n=240) will be randomly allocated to either the treatment arm (verum Coldamaris plus, 0.12% iota-carrageenan plus 0.04% Kappa-Carrageenan in 0.5% saline) or placebo (Coldamaris sine, saline 0.5%) arm. The study's primary objective is the prevention of COVID-19 infection, confirmed by PCR swab or documented seroconversion. Secondary objectives are to determine if carrageenan sprays reduce the clinical severity of COVID-19 and symptomatic acute respiratory infection of other aetiologies (non-SARS-CoV-2).

DETAILED DESCRIPTION:
Objectives:

The primary objective is to determine whether carrageenan nasal and throat sprays reduce the risk of COVID-19 infection.

The secondary objectives are:

1. To determine whether carrageenan nasal and throat spray reduces the severity and/or duration of COVID-19 infection;
2. To determine whether carrageenan nasal and throat spray reduces the risk of infection with other respiratory viruses
3. To determine whether carrageenan nasal and throat spray reduces the severity and/or duration of infection with other respiratory viruses
4. To determine the usability of carrageenan nasal and throat spray for long term prophylaxis against respiratory viruses
5. To determine the effect on of using the spray on quality adjusted life years and cost effectiveness

Study Design:

The study design consists of a double blind, randomised placebo-controlled trial. Of the 480 healthcare professionals recruited, 240 participants will be randomly allocated to each of either the treatment arm (verum Coldamaris plus i.e. Iota-carrageenan 0.12% plus 0.04% Kappa-Carrageenan in 0.5% saline) or placebo (Coldamaris sine i.e. 0.5% saline) arms. Participants will use the spray prophylactically into each nostril and throat three times per day for 8 weeks, during which time the participants will be invited to complete a daily symptom tracker questionnaire. COVID-19 infection during the trial period will be confirmed using viral PCR swabs (if symptomatic), SARS-CoV-2 serology at 14 days following onset of symptoms as well as trial entry and exit serology to detect asymptomatic infection during the study period.

Allocation to each group, treatment or placebo administration and data analysis will be blinded to both participant and investigator. The primary outcome measure will be acquisition of COVID-19 infection as confirmed by positive PCR swab taken at the time of symptoms or positive serology measured 2 weeks after symptom onset or seroconversion at the end of the trial (via trial entry and exit serology) to detect asymptomatic infection during the study period. Secondary outcome measured will include symptom types, severity and duration (recorded by the daily symptom tracker questionnaire), hospital admission and length of stay, oxygen saturation and radiological lung changes on admission, need for ventilatory support (oxygen therapy, CPAP, intubation & ventilation), haematological changes, intensive care admission and length of stay, mortality, subsequent familial/household COVID-19 infection and acquisition of non-COVID-19 upper respiratory tract infections.

Deliverables:

1. This trial will help us to determine whether carrageenan nasal sprays significantly affect the primary outcome measure of acquisition of COVID-19 infection as confirmed by positive PCR swab taken at the time of symptoms or positive serology measured 2 weeks after symptom onset or at the end of the study.
2. It will also determine the effect of carrageenan nasal sprays on secondary outcome measures which include types, severity and duration of symptoms, hospital admission and length of stay, need for ventilatory support and intensive care admission, mortality as well as familial or household COVID-19 infection and acquisition of other respiratory tract infections.
3. We will also investigate whether haematological changes (FBC, CRP, U&E, Ferritin, LFT, LDH, Clotting, D-dimer, FDP, Vitamin D level) and demographic questionnaire findings can offer a predictive value for acquiring COVID-19 infection or determining severity and/or duration of resultant infection.
4. To determine any associations between symptom severity and/or duration and prognosis in those with COVID-19.
5. Determine usability and acceptability of nasal and throat spray as prophylaxis and affect on quality adjusted life years and cost effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Study participants who have given informed consent, and received a copy of signed consent form prior to any study related procedures;
* Healthcare professionals (nurses, doctors, allied health professionals, health care assistants, operating department practitioners) working in Swansea Bay University Health Board initially as well as any other volunteers >18 years who have not previously tested positive for COVID19 or been vaccinated.
* Subjects agree to refrain from taking over the counter products intended to prevent, intervene in, or treat colds/flu, starting at study entry and continuing through week 10 of the study.

Exclusion Criteria:

Capacity, consent and conflicts of interest:

* The person lacks capacity;
* The subject is related to any study personnel or has any other close ties or conflicts of interest with the research team or the study sponsor;
* The subject has received any investigational drug or participated in a clinical trial within 4 weeks of entry to this study.
* Unable to complete the daily symptom tracker
* Unable to communicate in English or Welsh

Comorbidities:

* Known hypersensitivity or allergy to any component of the test product;
* Severe cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease, immune deficiency, autoimmune disease or a history or any current disease that is considered by the investigator as a reason for exclusion;
* Severe nasal septal deviation, nasal polyps or other non-infectious condition that could cause nasal obstruction;
* A history of any nasal or sinus surgery in the past that in the opinion of the investigator may influence the symptoms or spray administration;
* An unrelated infection that in the opinion of the investigator may influence symptoms (gastrointestinal infection, other viral diseases such as measles, mumps);

COVID-19 Status:

* Participants with proven COVID-19 infection (previous positive serology and/or viral PCR swab)
* Participants that have already received their vaccination or already booked in for their vaccination

Medications:

* Recent treatment of common cold that in the opinion of the investigator may influence symptoms (see Table 2)
* Participants taking any of the medications outlined in Table 2 during the trial period will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 infection | 9-12 months
  Acquisition of COVID-19 infection as confirmed by positive PCR swab taken at the time of symptom onset or positive serology measured 2 weeks after symptom onset or seroconversion at the end of the trial (via trial entry and exit serology) to detect asymptomatic infection during the study period

SECONDARY OUTCOMES:
Duration of COVID-19 infection | 9-12 months
  Time taken for all symptoms to resolve (days)
Hospitalisation due to COVD-19 infection | 9-12 months
  Length of hospital and intensive care stay (days)
Severity of COVID-19 infection | 9-12 months
  Morality rate
Quality of life of nasal spray use | 9-12 months
  Usability of spray and effect on cost and quality adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Zita M Jessop, MBBChir PhD, Principal Investigator — Swansea University
Locations (1):
- Joint Clinical Research Facility, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buck CB, Thompson CD, Roberts JN, Muller M, Lowy DR, Schiller JT. Carrageenan is a potent inhibitor of papillomavirus infection. PLoS Pathog. 2006 Jul;2(7):e69. doi: 10.1371/journal.ppat.0020069. PMID 16839203
- [Background] Eccles R, Meier C, Jawad M, Weinmullner R, Grassauer A, Prieschl-Grassauer E. Efficacy and safety of an antiviral Iota-Carrageenan nasal spray: a randomized, double-blind, placebo-controlled exploratory study in volunteers with early symptoms of the common cold. Respir Res. 2010 Aug 10;11(1):108. doi: 10.1186/1465-9921-11-108. PMID 20696083
- [Background] Eccles R, Winther B, Johnston SL, Robinson P, Trampisch M, Koelsch S. Efficacy and safety of iota-carrageenan nasal spray versus placebo in early treatment of the common cold in adults: the ICICC trial. Respir Res. 2015 Oct 5;16:121. doi: 10.1186/s12931-015-0281-8. PMID 26438038
- [Background] Gonzalez ME, Alarcon B, Carrasco L. Polysaccharides as antiviral agents: antiviral activity of carrageenan. Antimicrob Agents Chemother. 1987 Sep;31(9):1388-93. doi: 10.1128/AAC.31.9.1388. PMID 2823697
- [Background] Grassauer A, Weinmuellner R, Meier C, Pretsch A, Prieschl-Grassauer E, Unger H. Iota-Carrageenan is a potent inhibitor of rhinovirus infection. Virol J. 2008 Sep 26;5:107. doi: 10.1186/1743-422X-5-107. PMID 18817582
- [Background] Ludwig M, Enzenhofer E, Schneider S, Rauch M, Bodenteich A, Neumann K, Prieschl-Grassauer E, Grassauer A, Lion T, Mueller CA. Efficacy of a carrageenan nasal spray in patients with common cold: a randomized controlled trial. Respir Res. 2013 Nov 13;14(1):124. doi: 10.1186/1465-9921-14-124. PMID 24219370
- [Background] Leibbrandt A, Meier C, Konig-Schuster M, Weinmullner R, Kalthoff D, Pflugfelder B, Graf P, Frank-Gehrke B, Beer M, Fazekas T, Unger H, Prieschl-Grassauer E, Grassauer A. Iota-carrageenan is a potent inhibitor of influenza A virus infection. PLoS One. 2010 Dec 14;5(12):e14320. doi: 10.1371/journal.pone.0014320. PMID 21179403
- [Background] Shao Q, Guo Q, Xu Wp, Li Z, Zhao Tt. Specific Inhibitory Effect of kappa-Carrageenan Polysaccharide on Swine Pandemic 2009 H1N1 Influenza Virus. PLoS One. 2015 May 13;10(5):e0126577. doi: 10.1371/journal.pone.0126577. eCollection 2015. PMID 25969984
- [Derived] Jessop ZM, Gibson J, Lim JY, Jovic TH, Combellack E, Dobbs TD, Carter K, Hiles S, Islam S, Healy B, Humphreys I, Eccles R, Hutchings HA, Whitaker IS. A study protocol for a double-blind randomised placebo-controlled trial evaluating the efficacy of carrageenan nasal and throat spray for COVID-19 prophylaxis-ICE-COVID. Trials. 2022 Sep 15;23(1):782. doi: 10.1186/s13063-022-06685-z. PMID 36109791